CLINICAL TRIAL: NCT04288882
Title: Role of Balloon-Assisted Enteroscopy (BAE) in Diagnosis and Treatment of Small Intestinal Disorders
Brief Title: Role of Balloon-Assisted Enteroscopy (BAE) in Small Intestinal Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Doctor, Assiut University
Other Study IDs: Role of enteroscopy
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Role of Enteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Enteroscopy — Role of Balloon-Assisted Enteroscopy (BAE) in management of Small Intestinal Disorders

SUMMARY:
Overall Aim:

This study is designed to assess the role of ballon-assisted enteroscopy in the management of obscure small intestinal disorders in a tertiary-care center in Upper Eygpt.

Specific objectives:

1. Evaluate the technical success rate and causes of the procedure in our locality
2. Explore the value and safety of BAE in the diagnose and treatment of suspected small bowel diseases.
3. Assess patients' and endoscopists' satisfaction related to the procedure.
4. Define the indications, diagnostic yield and appropriatness of BAE in our center.
5. Determine the value of enteroscopy-obtained biopsy samples in the diagnosis.
6. Perform a cost analysis of BAE in relation to its diagnostic value/yield.
7. Report the therapeutic role of BAE in different small intestinal disorders.

DETAILED DESCRIPTION:
The small intestine is very essential for digestion and absorption and is presented between the stomach and large intestine. Because of its anatomical position, the small intestine was named as a "blind area" leading to difficulty in diagnosis of small bowel disease. The advant of ballon-assisted enteroscopy facilitates the management of the small bowel diseases. There are several causes of obscure small intestinal disorders, which are Angioectasia (20-55%), small bowel tumours (10-20%), Cameron erosions (5-15%), NSAID enteropathy (5%), Dieulafoy lesion (2-3%), Crohn's disease (2-10%), Coeliac disease( 2-5 %), Meckel's diverticulum (2-5%), duodenal varices (1-5%), gastric antral vascular ectasia (GAVE) (1-2%), Ectopic varices (1-2%), Portal hypertensive enteropathy 1-2% (but 60-70% in those with portal hypertension), Radiation enteritis (<1% ). Obscure gastrointestinal bleeding (OGIB) was the most common indication for enteroscopry and is defined as a bleeding from an unknown site after a negative evaluation of the GI tract with esophagogastroduodenoscopy (EGD) and ileocolonoscopy. OGIB represents about 5% of patients presenting with GI bleeding. OGIB isthe most common indication for enteroscopry, whatever the age groups, but the proportion of patients performing enteroscopy for OGIB was higher in elderly patients. Young patients were indicated for enteroscopy for other complains, such as abdominal pain, or suspicious small-bowel tumor. Egyptian study was done and identified that the source of OGIB in the small intestine represents 69.2%, with negative DBE ﬁndings in 30.8% and the most common lesions were angioectasias followed by GI tumours (30.8%, 19.2%, respectively).

ELIGIBILITY:
Inclusion Criteria:All male and female patients aged ≥18 - ≤80 year-old with suspected small intestinal disorders referred to the above Unit for BAE in the period between March 2020 till March 2022 inclusive irrespective of indication will be included in this study.

Exclusion Criteria:Those who are <18 years-old and >80 years-old, those with gastrointestinal obstruction, preganat ladies, and those who fail to provide consent will be excluded.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After obtaining the appropriate consents, data pertaining to clinical history, physical examination and baseline laboratory investigations (complete blood count, kidney function, coagulation profile) for all cases of obscure small intestinal disorders. CT abdomen, conventional upper GI endoscopy and colonoscopy in addition to other modalities as the CT scan and angiography will be done for every patient as appropriate.
  All patients will be subjected to the BAE if these modalities are negative. BAE will be performed in an outpatient or inpatient setting under general anesthesia, although some patients may require only conscious sedation. Most procedures will be performed through the mouth (antegrade), although the (retrograde) approach, through the rectum, may be done resorted to allow better access to suspected lesions in the lower part of the small bowel.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Role of Balloon-Assisted Enteroscopy (BAE) in Diagnosis and Treatment of Small Intestinal Disorders | baseline
  This study is designed to assess the role of ballon-assisted enteroscopy in the management of obscure small intestinal disorders in a tertiary-care center in Upper Eygpt.

REFERENCES:
- [Background] Hashimoto R, Nakahori M, Matsuda T. Impact of Urgent Double-Balloon Enteroscopy on the Short-Term and Long-Term Outcomes in Overt Small Bowel Bleeding. Dig Dis Sci. 2019 Oct;64(10):2933-2938. doi: 10.1007/s10620-019-05627-1. Epub 2019 Apr 17. PMID 30997580